CLINICAL TRIAL: NCT04859400
Title: Influence of a Home-based Nutrition and Exercise Program Including an Application for Monitoring on Quality of Life in Palliative Cancer Outpatients
Brief Title: Influence of a Home-based Nutrition and Exercise Program on Quality of Life of Palliative Cancer Outpatients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kantonsspital Winterthur KSW (Other)
Collaborators: Krebsforschung Schweiz, Bern, Switzerland (Other); Sponser Sport Food AG (Unknown); Leitwert GmbH (Unknown); SNAQ AG (Unknown); Cantonal Hospital of St. Gallen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2020-02992
Record Dates: First submitted 2021-04-08; First posted 2021-04-26 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Cancer, Gastrointestinal; Cancer, Lung; Malnutrition
Keywords: Cancer; Palliative; Application; Nutrition; Exercise
MeSH Terms: conditions — Gastrointestinal Neoplasms; Lung Neoplasms; Malnutrition; Neoplasms; Motor Activity | interventions — Leucine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): standardized nutritional program including a nutritional supplement
  standardized exercise program
  app for monitoring.
  Interventions: Dietary Supplement: Whey protein supplement high in leucine and β-hydroxy-β-methylbutyrate (HMB); Behavioral: Standardized nutritional program; Behavioral: Standardized exercise program
- Control (No Intervention): standard of care
  limited version of the app (e.g. without the "help" function).

INTERVENTIONS:
Dietary Supplement: Whey protein supplement high in leucine and β-hydroxy-β-methylbutyrate (HMB) — The whey protein supplement high in leucine and β-hydroxy-β-methylbutyrate (HMB) is ingested once daily, preferably either in the evening before going to bed or within two hours after having finished exercising.
  Arms: Intervention
Behavioral: Standardized nutritional program — During at least two personal counseling meetings with a dietician, the patient's diet is assessed and individual nutritional interventions - based on the personal needs and individual preferences of the patient - are developed. The overall goal is to optimize protein an energy intake.
  Arms: Intervention
Behavioral: Standardized exercise program — In at least two personal counseling meetings with a physiotherapist, the patient's individual training plan is compiled and agreed upon (mainly including strength, endurance and balance exercises). The patient then exercises at home and records the trainings with the app.
  Arms: Intervention

SUMMARY:
The main purpose of the study is to investigate whether a tailor-made nutritional and exercise program including home-based sessions and regular monitoring using an application on the smartphone is effective in improving Quality of Life in patients with advanced lung or gastrointestinal tract cancer.

DETAILED DESCRIPTION:
Cachexia is highly prevalent among cancer patients and has substantial impact on the Quality of Life (QoL) and the functional status of patients.Therefore, the main purpose of this study is to investigate whether a mainly home-based nutritional and exercise program including regular monitoring using an application on the smartphone is effective in improving QoL in patients with advanced lung or gastrointestinal tract cancer.

The study desing is a randomized, two-arm and multicenter international trial and advanced lung or gastrointestinal cancer patients not eligible for curative treatment make up the patient population.

Patients in the intervention group receive a nutrition and exercise program in combination with an electronic application for data collection and monitoring.

The nutritional program comprises an extensive nutritional assessment and an individual nutritional recommendation. In addition, patients receive a whey protein supplement high in leucine and β-hydroxy-β-methylbutyrate (HMB) to support an optimal protein intake in combination with physical activity. The nutritional situation is reassessed at 2 -3 weeks.

Exercise counselling includes at least two visits with an extensive first baseline assessment. On this basis, an individual training program for 12 weeks in a home-based setting is compiled, with mainly strength and endurance exercises. At week 2-3, the patient and the study physiotherapist have a follow-up meeting.

The application Swiss NutriAct is mainly used for data collection (nutritional, exercise and QoL data). Since the study coordinator, dietician and physiotherapist can see the information entered by the intervention group patients, they can contact patients and offer help regarding the nutrition and exercise program, where deemed appropriate. Vice versa, patients can use the help button to contact the study team to ask questions regarding the nutrition and exercise program.

Patients in the control group receive standard of care and a limited version of the application.

Both arms will be assessed at baseline (0 weeks), after the 12 weeks intervention phase and at a follow up assessment after 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Advanced lung or gastrointestinal cancer patients not eligible for curative treatment
* WHO performance status of ≤ 2
* Able to perform physical exercise estimated by the treating physician
* Estimated life expectancy of ≥ 6 months
* Patient must give written informed consent

Exclusion Criteria:

* Intake of supplements with high-dose branched-chain amino acids within one month
* Enteral (except oral nutritional supplements) and/or parenteral nutrition within one month
* History of ileus within previous month
* Milk protein allergy
* The patient cannot understand the trial-specific content due to linguistic, psychological or disease reasons
* Age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2021-06-07 (Actual); Primary Completion 2024-09-12 (Actual); Study Completion 2024-11-06 (Actual)

PRIMARY OUTCOMES:
QoL | 3 Months
  Questionnaire Functional Assessment of Cancer Therapy - General (FACT-G)

SECONDARY OUTCOMES:
Nutritional status | 3 months
  Body weight (in kg), used in combination with body height to calculate BMI (in kg/m2)
Nutritional status | 3 months
  Patient-generated subjective global assessment (PGSGA)
Nutritional status | 3 months
  Bioelectrical impedance analysis (BIA)
Nutritional status | 3 months
  Muscle mass: L3 image of computertomographic (CT) measurements taken in the context of standard cancer therapy (divided by height squared; in cm2/m2)
Nutritional status | 3 months
  Calf circumference (in cm)
Nutritional status | 3 months
  Sarcopenia screening questionnaire SARC-F
Physical function | 3 months
  Handgrip strength (in kg)
Physical function | 3 months
  60 s sit-to-stand test (number of stands)
Physical function | 3 months
  6 minute walk test (in m)
Energy- and protein intake | 3 months
  Data collected with application, Harris-Benedict formula
Fatigue | 3 months
  Questionnaire Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-Fatigue)
Clinical data | 3 months
  Physical performance status (WHO performance status, grade 0-5)
Clinical data | 3 months
  Tumor stadium
Clinical data | 3 months
  Adverse events grade 3 and 4
Clinical data | 3 months
  Serious adverse events
Clinical data | 3 months
  Unplanned hospital readmissions
Clinical data | 3 months
  Survival
Adherence to the nutritional and exercise program | 3 months
  According to data collected with application
Usability of the new application | 3 months
  Questionnaire mHealth App Usability (MAUQ)
Success of recruitment rate in comparison to former studies | Through study completion (24 months)
  Number of eligible patients, participants, rejections as compared to similar past studies

CONTACTS AND LOCATIONS:
Overall Officials: Christian Britschgi, PD Dr. med. Dr. phil, Principal Investigator — Kantonsspital Winterthur KSW
Locations (3):
- Klinikum Konstanz, Konstanz, Germany
- Switzerland (2):
  - Spital STS (Simmental-Thun-Saanenland) AG, Thun
  - Kantonsspital Winterthur, Winterthur

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data (IPD) with other researchers.